CLINICAL TRIAL: NCT05533060
Title: Clinical and Molecular Biological Data Collection and Analysis in Patients With Traumatic Brain Injury (TBI)
Brief Title: Clinical and Molecular Biological Data Collection and Analysis in Patients With TBI
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Chen, MD, PhD, Associate Clinical Professor, Supervisor, Shanghai 6th People's Hospital
Other Study IDs: 2022-KY-13(K)
Record Dates: First submitted 2022-09-06; First posted 2022-09-08 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; Molecular biomarkers; Single-cell sequencing; High-throughput sequencing
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — 1. Brain tissues removed by decompression in patients with traumatic brain injury (TBI)
  2. Cerebrospinal fluid (CSF)
  3. Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TBI group: patients with traumatic brain injury (TBI) treated surgically
  Interventions: Other: No intervention
- RN group: relatively normal (RN) participants including patients with other brain diseases, for example, gliomas, meningiomas, and schwannomas, treated surgically
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — patients in the groups are treated surgically and brain tissue, CSF, and blood samples, as well as clinical data, neuroimaging data are collected

SUMMARY:
Clinical evaluation is crucial in the clinical diagnosis, treatment, and prognosis prediction in patients with traumatic brain injury (TBI). However, the existing evaluation systems are not perfect, because many factors are not taken into account, for example, there is a lack of molecular diagnostic criteria for evaluating patients with TBI. We attempt to collect the patient's clinical data and combine it with neuroimaging, as well as molecular biomarkers generated by single-cell sequencing to assess their neurological status and outcome. The clinical and molecular data collection and analysis will be helpful to evaluate the patient's neurological condition and predict the patient's outcome more accurately.

DETAILED DESCRIPTION:
Specifically, eligible patients will be treated surgically. In one group, injured brain tissue removed during decompression and resection will be preserved in a tissue preservation solution. In another group, brain tissue in the surgical trajectory during surgical resection of the brain lesion (for example, gliomas, meningiomas, schwannomas) will be also preserved in the solution. Then these tissues will be analyzed through high-throughput single-cell sequencing and bioinformatics analysis. In order to obtain the most changed biomarkers, we will pick up the top 10 cell subgroups with 10 expression biomarkers in each subgroup to compare them with the results analyzed in the mice brain tissue. The target biomarkers will be validated in the cerebrospinal fluid (CSF) and blood in patients with TBI for the patient's neurological status evaluation and outcome prediction. At the same time, the patient's pre- and postoperative clinical data (including, gender, age, GCS score, pupil light reflection, CT results, etc) will also be collected. A regression model will be generated to estimate the relationship between the patient's neurological status and these independent variables. In addition, the association between a patient's prognosis and these factors will also be analyzed. ROC curve will be used to compare our regression model to the established GCS score scale and Marshall CT grading.

ELIGIBILITY:
Inclusion Criteria:

* CT/MRI confirmed TBI;
* The time from onset to the emergency room (ER ) within 12h;
* The systolic pressure (SBP) ≥ 90 mmHg;
* Patients willing to participate in this study with signed informed consent.

Exclusion Criteria:

* Patients who are not suitable for surgery (GCS score 3 points, dilated and fixed bilateral pupils, pregnant women, etc.);
* Pre-injury life expectancy ≤ 1 year (malignant tumor);
* Previous history of acute myocardial infarction, abnormal immune function, and blood-related diseases;
* without informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with traumatic brain injury (TBI) or other brain diseases (gliomas, meningiomas, schwannoma) who are treated surgically
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Accurate assessment of patients' neurological condition | 2022.09-2023.12
  Using a regression model to explore the relationship between a patient's neurological condition and clinical and molecular biological data

SECONDARY OUTCOMES:
Predicting patients' outcome accurately | 2022.09-2023.12
  Using a regression model to explore the relationship between a patient's prognosis and clinical and molecular biological data

CONTACTS AND LOCATIONS:
Overall Officials: Hengli Tian, MD, PhD, Study Director — Shanghai 6th People's Hospital
Locations (1):
- Shanghai 6th People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD could be available on from the central contact person with a reasonable request.